CLINICAL TRIAL: NCT01149135
Title: Randomized and Controlled Study of the Effects of Low Intensity 'Blue Light'in the Treatment of Seasonal Affective Disorder
Brief Title: Low Intensity 'Blue Light' Treatment of Seasonal Affective Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Ybe Meesters PhD, University Medical Center Groningen
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: METc 2008.184
Record Dates: First submitted 2010-06-22; First posted 2010-06-23 (Estimated); Last update posted 2011-08-10 (Estimated); Status verified 2008-10

CONDITIONS: Seasonal Affective Disorder
Keywords: Seasonal Affective Disorder; phototherapy; circadian rhythms; blue enriched light; melanopsin; low intensity
MeSH Terms: conditions — Seasonal Affective Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard light treatment (Active Comparator): standard light treatment 5000K; 10 000 lux
  Interventions: Device: standard light treatment
- blue enriched light (Experimental): Blue enriched light with a low intensity (750 lux)
  Interventions: Device: Blue enriched light with a low intensity

INTERVENTIONS:
Device: Blue enriched light with a low intensity — 30 minutes in the morning, 750 lux
  Other Names: Blue enriched light treatment; Philips energy light HF 3309, 2 lamps PLL36 W 17000 K
  Arms: blue enriched light
Device: standard light treatment — standard light treatment, 30 minutes, 10 000 lux
  Other Names: Philips Energylight HF 3309, 2 lamps PLL36 W, color 5000K, 10 000 lux
  Arms: Standard light treatment

SUMMARY:
One of the most frequently investigated hypothesis of the pathophysiology underlying Seasonal Affective Disorder(SAD) or so called winter depression is a disturbance of circadian rhythms. Since the circadian system is especially sensitive for the blue portion of the light spectrum, a new light therapy device with more blue light (blue enriched polychromatic light) was tested for its efficacy to treat SAD. In chronobiological terms this light is hypothesized to be more potent in inducing non-visual effects. In the present study fluorescent tubes that emit a high portion of short wavelength light on top of the normal wavelengths are tested for its superiority in treating SAD. This blue-enriched light (colour temperature 17000 ºK) is compared to standard light treatment (5000 º K) in SAD patients.,In a earlier study it was shown that the therapeutic effect of blue enriched light were equal to standard light treatment using light in both conditions with an intensity of 10 000 lux. In the present study, blue enriched light with an intensity of 750 lux was used, because of the possible saturation effect in the former study. The investigators hypothesise that blue- enriched light with a low intensity improve the therapeutic effects of light treatment leading to a higher response or the same response in a shorter time schedule compared to standard light treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65
* Diagnose of Seasonal Affective Disorder, winter type according to DSM-IV SIGH SAD rating Higher then or equal to 18 on day 1
* No other treatments for mood disorder during the study
* Stay in the Netherlands during the study

Exclusion Criteria:

* Other axis-I disorders according to the DSM-IV
* Acute suicide risk
* Use of psychotropic drugs or photosensitizing drugs
* No other treatments for mood disorder during the study
* Diabetes or epilepsy
* Regular shift work

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2008-10; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
SIGH-SAD | weekly
  Structured Interview Guide of the Hamilton Depression Scale, seasonal affective disorder version